CLINICAL TRIAL: NCT04155970
Title: In Patients With Acute Non-specific Low Back Pain, do Lumbar Inter-vertebral Motion Variables Change Following a Course of Manual Therapy: A Feasibility Study
Brief Title: The Biomechanical Effects of Manual Therapy - A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: AECC University College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Version 1.0
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain, Mechanical
Keywords: Manual Therapy; Fluoroscope; Mechanics; Kinematics
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is blinded as to which intervention each participant received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy Arm (Experimental): The group will receive manual therapy, as well as an evidence-informed home management booklet.
  Interventions: Other: Manual therapy; Other: Evidence-informed home management booklet
- Non-Manual Therapy Arm (Experimental): The group will receive an evidence-informed home management booklet only.
  Interventions: Other: Evidence-informed home management booklet

INTERVENTIONS:
Other: Manual therapy — Manual therapy, which includes spinal manipulation; spinal mobilisation; light massage; and trigger point therapy.
  Arms: Manual Therapy Arm
Other: Evidence-informed home management booklet — The home management booklet includes advice on posture, over the counter pain medication, cold and heat packs. The booklet also includes a section on patient reassurance and where to seek help from a medical professional in an emergency.
  Other Names: Low back pain self help booklet

SUMMARY:
The aim of this study is to determine the feasibility of conducting a full-scale trial to explore if there is a change in intervertebral movement following a course of manual therapy in patients with acute non-specific low back pain (NSLBP).

Research Questions:

1. In patients with acute NSLBP, does lumbar intervertebral movement change following a course of manual therapy?
2. In patients with acute NSLBP, do those who respond to manual therapy (established by patient reported outcomes measures) have different intervertebral movement to those who do not?

DETAILED DESCRIPTION:
Non-specific low back pain (NSLBP) is a leading cause of disability and work-days lost worldwide. Yet, in most cases we do not know the specific cause. It is thought to be due to abnormal movement between the spinal bones (vertebrae). The investigators can now measure movement between vertebrae using low-dose quantitative fluoroscopy (QF), or motion x-ray videos. QF is a reliable method of measuring spinal movement which is non-invasive and does not expose the patient to a lot of radiation. In this study, QF will be used as a measuring tool to measure spinal movement in patients with acute NSLBP before manual therapy versus after manual therapy to explore if there is a change in spinal movement. Research suggests that some patients respond to manual therapy and some do not, a secondary question in this study is to explore if there are differences in spinal movement between those who respond to manual therapy (measured using pain and disability questionnaires) and those who do not.

This study is a feasibility study to determine whether the study can be carried out as a full-scale trial. Participants will be recruited from the AECC University College (AECC UC) Clinic. Following an examination, patients with acute low back pain, and who are eligible for the study will be invited to join. Participants will proceed with initial measurements which include validated questionnaires and QF. Following these measurements participants will be randomised into two groups, each containing 15 participants. Both groups will receive an evidence-informed home management booklet, the manual therapy group will receive five manual therapy treatments in two weeks. Participants will return for follow-up measurements two weeks after baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute non-specific low back pain (NSLBP), without leg pain, of at least 2 weeks duration, but no more than 4 weeks duration
* Patients between the ages of 18 and 65

Exclusion Criteria:

* Patients who cannot understand written English and unable to provide full informed consent.
* Patients who are currently involved in another research study
* Patients with a BMI over 30 (less likely to obtain the required information from the images)
* Pregnancy or potentially pregnant
* Previous ionising radiation exposure within the last 6 months greater than 8mSv.
* Previous lumbar spine surgery, as well as recent abdominal or pelvic surgery (within the last 12 months).
* Scoliosis or positive Adams forward Bending Test for Scoliosis.
* Diagnosed Osteoporosis (Bone Density Scan)
* Patients with a numeric pain scale of 8 or more, or 2 or less, taken at the New Patient Examination Appointment.
* Manual therapy already received for this episode of NSLBP
* Litigation or compensation pending
* Diagnosis of depression (by a medical doctor) within the last 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Ratio of presenting patients and eligible patients | 1 year
  Ratio of the number of patients seeking care for acute non-specific low back pain vs. number of eligible patients (according to eligibility criteria)
Ratio of patients approached vs. number of participants who consent to trial | 1 year
  Rate of conversion from number of patients approached (who are eligible for the trial) to number of participants who consent to be a part of the trial.
Incidence of participant withdrawal | 1 year
  Total participant number in the trial vs. number of participants who withdraw from the trial (where the participant withdraws from the trial)
Incidence of participant being withdrawn | 1 year
  Total participant number in the trial vs. number of participants who have been withdraw from the trial (where the practitioner withdraws the participant from the trial)
Participant compliance in arm one | 1 year
  Ratio of total participants in arm one vs. number of participants who were non-compliant with the intervention (in arm one)
Participant compliance in arm two | 1 year
  Ratio of total participants in arm two vs. number of participants who were non-compliant with the intervention (in arm two)
Number of participants who experienced adverse or serious adverse events | 1 year
  Ratio of total number of participants (in both groups) vs. serious adverse events, as well as adverse events.

SECONDARY OUTCOMES:
Bournemouth Questionnaire | 2 weeks
  Baseline and follow up Bournemouth Questionnaire scores. Scale data from 0 - 70, where 0 is the best outcome and 70 is the worst outcome. Minimally Important Change = 26.
Roland Morris Disability Questionnaire - 24 | 2 weeks
  Baseline and follow up Roland Morris Disability Questionnaire - 24. Scale data from 0 - 24, where 0 is the best outcome and 24 is the worst outcome. Minimally Important Change = 5.
Inter-vertebral range of angular motion | 2 weeks
  Baseline and follow up measurement taken from Quantitative Fluoroscopy (QF). QF systems combines fluoroscopy, with a computer-based process which tracks the vertebrae motion and calculates inter-vertebral movement variables.
  Inter-vertebral range of angular motion is scale data measured in degrees.
Sagittal translation | 2 weeks
  Baseline and follow up measurement taken from Quantitative Fluoroscopy (QF). Sagittal translation is scale data measured in millimetres.
Laxity | 2 weeks
  Baseline and follow up measurement taken from Quantitative Fluoroscopy (QF). Laxity is scale data and represents initial attainment rate.
Anterior disc height | 2 weeks
  Baseline and follow up measurement taken from Quantitative Fluoroscopy (QF). Anterior disc height is scale data measured in millimetres.
Motion Sharing Inequality (MSI) | 2 weeks
  Baseline and follow up measurement taken from Quantitative Fluoroscopy (QF). MSI is scale data and calculated as the average of the maximum distances between levels (L2-L5) at all data points.
Motion Sharing Variability (MSV) | 2 weeks
  Baseline and follow up measurement taken from Quantitative Fluoroscopy (QF). MSV is scale data and calculated as the square root of the variance between levels (L2-L5) at all data points.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Sewell, Study Chair — Head of Department - Design & Engineering
Locations (1):
- Bournemouth University, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the project is complete, the final anonymised dataset captured during the study will be uploaded to BORDaR (Bournemouth Online Research Data Repository). This is in the interest of open data sharing.
Supporting Information: CSR
Time Frame: An embargo will be placed on the final dataset until the study (and PhD) is complete and the results of the study have been published. In the interest of open data sharing, the data will be available indefinitely.
Access Criteria: Request for anonymised dataset will need to be submitted through BORDaR (Bournemouth Online Research Data Repository)
URL: http://bordar.bournemouth.ac.uk/